CLINICAL TRIAL: NCT04191122
Title: Community Outpatient Psychotherapy Engagement Service for Self-harm (COPESS): A Feasibility Study
Brief Title: Community Outpatient Psychotherapy Engagement Service for Self-harm
Acronym: COPESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Liverpool (Other); University of Manchester (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Pooja Saini, Senior Lecturer, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIHR200543
Record Dates: First submitted 2019-11-05; First posted 2019-12-09 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Self-Harm; Depression
Keywords: Primary care; Community settings
MeSH Terms: conditions — Self-Injurious Behavior; Depression

STUDY DESIGN:
Intervention Model Description: COPES is a brief (4 + 1 sessions, 50 minutes) psychotherapy based on psychodynamic and cognitive analytic principles that was developed to help those struggling with SH and depression. COPES is designed to be brief and accessible and involves working collaboratively with a client to try and identify patterns or conflicts in emotional experiences and interpersonal relationships, linked to depressed mood and acts of SH. The therapist works with the client to build a shared map or understanding of these experiences. A goal of therapy is to work towards a small number of specific "exits", representing helpful steps the client might make to improve their difficulties. Therapy would take place either in the participant's home or in a community setting (e.g. health centre or clinic) depending on preference.
  Safety for the therapist and/or mobility for the patient will be reviewed throughout the recruitment period. Participants in the COPES arm of the trial will also receive TAU.
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomized to receive COPES plus TAU or TAU via a random sequence generation computer algorithm within STATA to generate (stratified) randomised (block) allocations. Randomisation will be carried out by the study statistician using an independent computerised randomisation system with a randomly sized block design with block sizes of 2, 4 and 6. The study population will be stratified for those receiving TAU and those receiving COPES plus TAU. Researchers completing study assessments will be masked to treatment allocation, facilitated by briefing members of the research team and participants on the need to avoid disclosure of treatment details. The trial will follow an Intent-To-Treat (ITT) protocol. Attrition and reasons for drop-out will be recorded where possible. Guidance will be sought from the patient advisory group on how to manage and minimise attrition over the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPESS and Treatment as usual (Active Comparator): COPES is a brief (4 + 1 sessions, 50 minutes) psychotherapy based on psychodynamic and cognitive analytic principles that was developed to help those struggling with SH and depression. COPES is designed to be brief and accessible, and involves working collaboratively with a client to try and identify patterns or conflicts in emotional experiences and interpersonal relationships, linked to depressed mood and acts of SH. The therapist works with the client to build a shared map or understanding of these experiences. A goal of therapy is to work towards a small number of specific "exits", representing helpful steps the client might make to improve their difficulties. Therapy would take place either in the participant's home or in a community setting (e.g. health centre or clinic) depending on preference.
  Safety for the therapist and/or mobility for the patient will be reviewed throughout the recruitment period. Participants in the COPES arm of the trial will also receive TAU.
  Interventions: Other: COPESS
- Treatment as usual only (No Intervention): The control group will receive Treatment-as usual (TAU), defined as the standard care provided to individuals struggling with self-harm (SH) as detailed within the 'Managing SH in primary care' NICE guidelines. These include: an initial comprehensive psychosocial assessment of skills and risks; co-production of a care and risk management care plan, which should include harm reduction plans, the need for between 3 and 12 sessions of psychological intervention as well as treatment for associated mental health conditions. Primary care practices in the control arm will be asked to provide information on what constitutes TAU within their organisation. This trial may enhance TAU as researchers will provide details of NICE guidance to GP practices that may not currently be following these guidelines. We will collect data regarding the acceptability of TAU for SH offered by GPs within both treatment arms.

INTERVENTIONS:
Other: COPESS — The intervention includes brief psychotherapy to be delivered within primary care settings
  Other Names: Community Outpatients Psychotherapy Engagement Service for Self-harm
  Arms: COPESS and Treatment as usual

SUMMARY:
Background: Self-harm (SH) is any act of intentional self-injury or self-poisoning, with or without the intention to die. People who SH are at high risk for future suicide and often suffer considerable emotional distress. Depression is common among people who SH and may be an underlying driver of self-harm behaviour. Treating depression in people who SH has the potential to reduce the risk of further SH and suicide. Self-harm is often repeated, and risk of repetition is highest immediately after an act of self-harm. Readily accessible brief talking therapies show promise in helping people who SH, but further evaluation of these approaches is needed. The Community Outpatient Psychological Engagement Service for Self-Harm (COPESS) is a brief talking therapy intervention for depression and self-harm. This intervention was shown to be feasible and acceptable in hospital emergency department settings, but accessibility was limited; thus, the investigators wish to develop and test a community-based version of this intervention. The COPESS project moves this therapy into a community setting, thereby increasing the number of people who can be helped, especially those in hard-to-reach groups and from disadvantaged areas.

Aim: To assess the feasibility of conducting a trial of the COPESS intervention in a community setting, for people with depression who self-harm, in relation to participant recruitment and retention. Therapy, acceptability and safety of the intervention will also be assessed.

Methods: Using a Single Blind Randomised Control Trial (RCT) design, the investigators will recruit a sample of n=60 participants with a history of SH within the last six months, who are also currently depressed. Recruitment will take place via GP practices for patients who: 1) seek consultation for self-harm; 2) have consulted for self-harm in the previous 6 months (determined by GPs' search of their own data-systems); or 3) self-refer via their GP. Following baseline assessment participants will be randomly allocated to either receive COPESS plus Treatment as Usual [TAU; n = 30)] or TAU alone (n=30). Follow-up assessments will take place at one, two and three months. Recruitment rates, attrition and data completeness will be monitored. Qualitative interviews with participants and stakeholders will further investigate feasibility.

DETAILED DESCRIPTION:
Design A mixed-method evaluation of a single-blind randomised controlled trial (RCT) will determine the acceptability and safety of the COPES intervention, in preparation for a future large-scale trial of the efficacy of COPES for depression in people who SH. People who have depression and SH in the community will be randomised to receive either COPES plus treatment-as-usual (TAU) or TAU alone.

Recruitment rates and power calculations This study is intended as a preliminary evaluation of the feasibility of conducting a future large-scale RCT of the COPES intervention. As, the investigators are not conducting any hypothesis testing of effectiveness, or estimation of prevalence (other than attrition) a formal power calculation is not appropriate. A recruitment target of n=60 (n=30 per trial arm) will be used. This is a common and realistic recruitment target for feasibility trials, and will allow adequate precision in estimating rates relevant to trial outcomes (e.g. attrition, adverse events). This will allow an overall attrition rate of 30% to be estimated with 95% confidence intervals of +/- 12% or, 16% for a single arm. This sample size is adequate for estimating relevant analysis parameters, such as the standard deviation of effects, which are needed for determining the feasibility of a later efficacy trial. To avoid high attrition rates, the investigators will keep participants engaged via text and/or telephone reminders. The previous pilot of HOPE within the ED achieved an average recruitment of nine eligible referrals each month. Sixty-one percent of participants engaged with the therapy and attended at least one session. Rates of attendance for SH at GP practices and walk-in centres in the Liverpool area have been estimated at 70 per month. Based on these figures a recruitment rate of 3 to 4 participants each month with a goal of n=60 participants overall is achievable.

Research Sites The research will take place in Liverpool, in the North West of England. The North West has particularly high rates of SH. Between April 2011 and March 2014, there were 16,405 presentations for deliberate SH to emergency departments within Merseyside and Cheshire. Liverpool local authority had one of the highest number of attendances for SH in this area (15%, n = 2,489). Therefore, Liverpool provides a good location for undertaking work on SH.

Recruitment of GP Practices Lead GPs and/or practice managers at practices identified as suitable for inclusion in the COPES study will be invited to take part in writing. Invitation packs will be given by GPs and followed up by a telephone/skype/face time/face-to-face contact from a member of the research team to ascertain level of interest, and if appropriate, to arrange a meeting to discuss the study in more detail. The Clinical Research Network (CRN) will assist with recruitment of GP practices and have provided a letter of support (see Appendix B). Clinicians will be briefed on the COPES trial and provided with guidance on referring patients in to the study. To assist recruitment, clinicians will be provided with a brief screening checklist to help identify patients where depression-linked SH may be a concern.

ELIGIBILITY:
Inclusion Criteria:

* Recent episode of SH (in the past six months, self-reported)
* A score of 14 or greater on the Beck Depression Inventory-II (BDI-II) corresponding to the BDI-II score where 14-19 = mild depression, 20-28 = moderate depression, >28 = severe depression
* Aged 16 years and over (SH is especially prevalent in adolescents and young adults and often this transitional age is neglected. This study will be offering at least TAU which young people may not otherwise access. To leave 16-18 year olds out of this study may be unethical and guidance from the British Psychological Society states that people aged 16 years and over can give informed consent)
* Help-seeking, defined as attendance at GP practices or self-referral into the trial

Exclusion Criteria:

* Non-English speaking
* Diagnosed with an intellectual disability as determined by review of clinical notes - the therapy has not yet been adapted for working with this population
* Experiencing severe problems with addiction to alcohol or illicit drugs
* Actively suicidal or psychotic and/or severely depressed and unresponsive to treatment as judged by clinical team
* Unable or unwilling to give written informed consent to participate in the study
* Currently receiving talking therapy for SH

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention assessed by the number of therapy sessions completed by participants in the intervention arm. | 2 years
  The proportion of patients who complete all agreed sessions of therapy will be recorded (> 60% excellent. 40-60% acceptable; less than 40% not acceptable). Analysis of data from semi-structured interviews with participants, who did and did not complete the therapy, and therapists who delivered the therapy.
Incidence of Treatment-Emergent Adverse Events as assessed by the adverse experiences in psychotherapy self-reported measure | 2 years
  The Adverse Experiences in Psychotherapy (AEP) self-report measure will identify adverse experiences liable to occur within psychological therapy. Safety will be assessed as part of routine monitoring of Serious Adverse Events (SAEs). Hospitalisation for any reason, medically serious acts of SH and suicidal crises (defined as participant having a plan and intent to make an imminent suicide attempt) will be regarded as SAEs. Where these occur, a review will take place to assess the plausibility of the SAE being due to the intervention. The occurrence of SAE and the results of the review process will be documented. In cases where SAE are potentially linked to the trial, withdrawal of participants, halting or terminating the trial will be considered as required.
Feasibility of the intervention assessed by the number of assessments completed by participants in the intervention arm | 2 years
  We will collect data on the amount of missing data on completed assessments

SECONDARY OUTCOMES:
Beck Depression Inventory-II: Depressive symptoms | 2 years
  Beck Depression Inventory-II - corresponding to the BDI-II score where 14-19 = mild depression, 20-28 = moderate depression, >28 = severe depression
Frequency and severity of self-harm ideation and behaviour using the Self-Injurious Thoughts and Behaviours Interview - short form (SITBI) which is a structured interview | 2 years
  Self-Injurious Thoughts and Behaviours Interview includes both quantitative and qualitative items that assess the presence, frequency, and characteristics of a wide range of self-injurious thoughts and behaviours, including suicidal ideation, suicide plans, suicide gestures, suicide attempts, and nonsuicidal self-injury
Frequency and intensity of SH urges over the preceding week using the Alexian Brothers Urge to Self-Injure Scale (ABUSI) to assess the frequency, intensity, and duration of the urge to self-injure. | 2 years
  Alexian Brothers Urge to Self-Injure Scale (ABUSI) is a uni-dimensional measure of the severity of the urge to self-injure and demonstrates high internal consistency and test-retest reliability. Responses are on a 7-point scale with a maximum total score of 30 and higher scores reflecting more intense urges to self-injure.
Emotion regulation will be measured using the emotion regulation questionnaire that consists of 10 items capturing two specific emotion regulation strategies, cognitive reappraisal and expressive suppression. | 2 years
  The Emotion Regulation Questionnaire uses a 7-point Likert scale, where 1 means "strongly disagree", 4 "neutral", and 7 means "strongly agree". The higher the scores the greater the use of the emotion regulation strategy.
Clinical Outcomes in Routine Evaluation (CORE-10) | 2 years
  Clinical Outcomes in Routine Evaluation that is used within clinical health settings. The measure has 6 high intensity/severity and 4 low intensity/severity items. Higher scores indicate higher levels of general psychological distress, where a total score of 11 or above is within the clinically significant range and scores above 13 likely indicated depression.
Help-seeking questionnaires using the The General Help-Seeking Questionnaire (GHSQ) and The Actual Help Seeking Questionnaire (AHSQ) to assess intentions to seek help from different sources and for different problems. | 2 years
  The General Help-Seeking Questionnaire (GHSQ) and The Actual Help Seeking Questionnaire (AHSQ). For these measures participants respond to each problem-type by rating their help-seeking intentions on a 7-point scale ranging from 1 ("extremely unlikely") to 7 ("extremely likely") for each help source option including "no one." Higher scores indicate higher intentions.
The Helping Relationship Questionnaire (HRQ) measures the patient's perspective of the therapist-patient relationship via an 11 self-report items. | 2 years
  Items for the HRQ are rated on a 6-point likert scale, ranging from -3 ("Strongly feel it is not true") to +3 ("Strongly feel it is true"). Total scores, computed by summing all items, range from -33 to 33, with higher total scores reflecting greater therapeutic alliance.
Demographic characteristics | 2 years
  Age, sex, ethnicity, education, employment, social deprivation, and clinical history will be recorded at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Saini, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Brownlow Medical Group, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No need to make data available to other researchers

REFERENCES:
- [Derived] Saini P, Hunt A, Clements C, Gabbay M, Mills C, Kvamme-Mitchell K, Tahir N, Mulholland H, Kullu C, Hann M, Duarte R, Murphy A, Guthrie E, Taylor P. Feasibility and acceptability of the Community Outpatient Psychotherapy Engagement Service for Self-harm (COPESS): randomised controlled trial. BJPsych Open. 2025 Aug 20;11(5):e190. doi: 10.1192/bjo.2025.10780. PMID 40831028
- [Derived] Saini P, Hunt A, Taylor P, Mills C, Clements C, Mulholland H, Kullu C, Hann M, Duarte R, Mattocks F, Guthrie E, Gabbay M. Community Outpatient Psychotherapy Engagement Service for Self-harm (COPESS): a feasibility trial protocol. Pilot Feasibility Stud. 2021 Aug 27;7(1):165. doi: 10.1186/s40814-021-00902-3. PMID 34452642
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617